CLINICAL TRIAL: NCT05414799
Title: Effect of Figure Eight Vision Exercise Combined With Chin Nodding and Neck Stretching Exercises on Computer Vision Syndrome
Brief Title: Effect of Exercises on Computer Vision Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ibrahim 462-21
Record Dates: First submitted 2022-05-11; First posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Neck Pain; Dry Eye Syndromes; Head Pain; Eye Strain; Asthenopia; Computer Vision Syndrome
Keywords: Computer vision syndrome; Digital eye strain; visual display terminal
MeSH Terms: conditions — Neck Pain; Dry Eye Syndromes; Headache; Asthenopia

STUDY DESIGN:
Intervention Model Description: The study included two groups i.e. experimental and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): in control group,33 participants (17=male, 16=female) performed figure eight vision exercise for 30 seconds once a day for 4 to 5 days per week for total duration of 4 week.
  Interventions: Other: figure eight vision exercise
- Experimental Group (Experimental): in experimental group, 33 participants (17=male, 16=female) performed figure eight vision exercise for 30 seconds followed by chin nodding for 20 second and followed by self neck stretching for 20 seconds. All the exercises are performed once a day for 4 to 5 days per week for total duration of 4 week.
  Interventions: Other: figure eight vision exercise; Other: chin nodding; Other: neck stretching

INTERVENTIONS:
Other: figure eight vision exercise — figure 8 vision exercise is performed in sitting position focus on a point 10 feet away, trace an imaginary horizontally figure 8 with eyes. keep tracing figure eight.
Other: chin nodding — chin nodding performed in sitting for keeping head placed straight over spine, place finger on chin and tuck-in the chin while head straight back until a stretch is felt at base of head.
  Arms: Experimental Group
Other: neck stretching — trapezius : neck flexion with opposite side bending and same side rotation for both sides.
  sternocleidomastoid : neck extension with opposite side bending and same side rotation for both sides.
  Arms: Experimental Group

SUMMARY:
Computer vision syndrome characterized as a complex of eye and vision problem related with activities which increase stress for close to vision. It includes a group of visual symptoms which occur from the extended viewing of the digital screen, when the demands of the task exceed the abilities of the viewer. Computer vision syndrome is an umbrella term that envelops many eye and environment-related problem that happen when the viewing need of the task increase the visual capability of the computer user which cause inefficacy to focus appropriately on computer images. Computer vision syndrome is also known as Digital Eye Strain.

DETAILED DESCRIPTION:
The continuous pandemic of COVID-19 has caused huge pressure in the medical services framework and adjusted the everyday way of life of normal individuals. Episodes of lockdown and social distancing have cut face to face connections, schooling, and working. During the lockdown time frame, individuals have depended on computers for data and entertainment, prompt a higher hazard to promote computer vision syndrome. Up to 90% of computer users whose spend 3 hours a day in front of computer screen suffers from computer vision syndrome.

Computer vision syndrome symptoms include blurred vision, headaches, dry eye (Tearing), eye redness, burning eye sensation, neck and shoulder pain. Posture problem most commonly seen in computer users. Screen radiation is not good for eye and due to screen radiation eye muscle fatigue occurs and static posture causes neck muscle fatigue. In Computer vision syndrome, we guide the participate to follow preventive measures for example, use of antiglare filter, self-neck muscle stretching, keep the distance between eye and screen is approximately between 40 and 76 cm, Proper sleep, antiglare glasses, proper lightning, ergonomics positioning of computer monitor and taking breaks during work may help to avoid Computer vision syndrome related symptoms i.e. Neck and shoulder pain, Eye Redness, Blurred vision, dry eye (tearing), Headache, burning eye sensation.From this study, Participants become aware of the importance of neck stretching exercise during computer usage and distance from screen.

Factor contributing in Computer vision syndrome include low screen brightness, no of hours of use per day, sitting position, position of screen, improper viewing distance, improper viewing angle, ocular diseases, medical diseases and aging and environment, imbalance of light between the computer screen and the surrounding.

Computer vision syndrome (CVS) is the main world related problem of the 21st century and its side effects influence almost around 70% of all computer users. All around the world, Computer vision syndrome is one of the public health problems and decrease usefulness at work increased error rate, reduce job satisfaction and impair visual capacities. Given the low accessibility and uses of personal defensive instrument, the high responsibility and the restricted break time while work with computer in developing countries, the burden of Computer vision syndrome is very high.

In the current quick time of innovation, our lives have become subject to computer utilization and limitless admittance to electronic devices, whether it is connected with our work, in instructive organizations, or for entertainment purposes. The proceeded and uncontrolled use has represented a threat to our wellbeing and a raised gamble for Computer Vision Syndrome (CVS). The greater part of these manifestations is connected with eye vision, eye muscles, light awareness, outer muscle framework and other general body symptoms. Around 64%-90% of individuals experience these side effects because of abuse and aimless utilization of computers. The frequency of new cases every year mounts to a million.

Computer vision syndrome is common phenomena amongst computer users. Computers have become necessary part of modern life. Now a day's computer is used in every field of work and everything converts hard to soft so computer users increase Computers are now extensively used in schools and at home as well. With increased popularity of notebooks, use of digital devices is no longer only limited to desktops. People use computer for work, web surfing, social networking and playing video games. In this techno-age, children as young as two years are given touch screen devices like iPads to play and learn with. Professional video game players in South Korea are known to spend as long as 18 hours per day in front of their screens at a stretch.

The American Optometric Association defines computer vision syndrome as a group of eye and vision-related problems that occur due to prolonged computer usage.

In current life today, it is assessed that worldwide around 60 million individuals suffer from computer vision syndrome, including kids and understudies are unfortunately acclimated with utilize the computerize screen and computer for extremely extended period of time. What make things worse are the new bad behavior patterns of the school and college students to study their subject using the computer rather than the book studies. The use of the internet which was now also increasingly popular causes workers to spend time in front of the computer at least 3 hours per day. The benefits gained from the use of computers were very numerous but not everyone was aware of the problems caused when using a computer, especially if working at the computer for too long and continuously.The rapid development of technology makes computers as a tool that facilitates work quickly and efficiently. Almost all fields of work today use computers as a tool to facilitate their work, there were around 100 million people use

ELIGIBILITY:
Inclusion Criteria:

* individuals who have been working on computer for at least 2 years for 3 hours per day.

Exclusion Criteria:

* any individual diagnosed with head injury, head trauma, tumor, craniotomy, congenital eye disease and any other visual deficits like cataract and retinopathy.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-06-11 (Estimated); Study Completion 2022-06-12 (Estimated)

PRIMARY OUTCOMES:
self administered questionnaire | 4 weeks
  self administered questionnaire is used to asses computer vision symptoms that comprises of six symptoms that are headache, blurred vision, burning eye sensation, dry eyes, eye redness and neck and shoulder pain with severity of mild, moderate and severe.
computer vision syndrome level instrument | 4 weeks
  It is used to assess symptoms and associated factors of computer vision syndrome and comprises of 10 questions.The scoring of questionnaire is as 0= never, 1=sometime and 2=always.The reliability of questionnaire is 0.986.

CONTACTS AND LOCATIONS:
Overall Officials: Ibraheem Zafar, MS-CPT, Principal Investigator — Shifa tameer e millat university Islamabad
Locations (1):
- Shifa tameer e millat university, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turkistani AN, Al-Romaih A, Alrayes MM, Al Ojan A, Al-Issawi W. Computer vision syndrome among Saudi population: An evaluation of prevalence and risk factors. J Family Med Prim Care. 2021 Jun;10(6):2313-2318. doi: 10.4103/jfmpc.jfmpc_2466_20. Epub 2021 Jul 2. PMID 34322430
- [Background] Al Tawil L, Aldokhayel S, Zeitouni L, Qadoumi T, Hussein S, Ahamed SS. Prevalence of self-reported computer vision syndrome symptoms and its associated factors among university students. Eur J Ophthalmol. 2020 Jan;30(1):189-195. doi: 10.1177/1120672118815110. Epub 2018 Nov 26. PMID 30474390
- [Background] Assefa NL, Weldemichael DZ, Alemu HW, Anbesse DH. Prevalence and associated factors of computer vision syndrome among bank workers in Gondar City, northwest Ethiopia, 2015. Clin Optom (Auckl). 2017 Apr 10;9:67-76. doi: 10.2147/OPTO.S126366. eCollection 2017. PMID 30214362
- [Background] Galindo-Romero C, Ruiz-Porras A, Garcia-Ayuso D, Di Pierdomenico J, Sobrado-Calvo P, Valiente-Soriano FJ. Computer Vision Syndrome in the Spanish Population during the COVID-19 Lockdown. Optom Vis Sci. 2021 Nov 1;98(11):1255-1262. doi: 10.1097/OPX.0000000000001794. PMID 34510149
- [Background] Wang L, Wei X, Deng Y. Computer Vision Syndrome During SARS-CoV-2 Outbreak in University Students: A Comparison Between Online Courses and Classroom Lectures. Front Public Health. 2021 Jul 8;9:696036. doi: 10.3389/fpubh.2021.696036. eCollection 2021. PMID 34307289
- [Background] Kim AD, Muntz A, Lee J, Wang MTM, Craig JP. Therapeutic benefits of blinking exercises in dry eye disease. Cont Lens Anterior Eye. 2021 Jun;44(3):101329. doi: 10.1016/j.clae.2020.04.014. Epub 2020 May 12. PMID 32409236
- [Background] Segui Mdel M, Cabrero-Garcia J, Crespo A, Verdu J, Ronda E. A reliable and valid questionnaire was developed to measure computer vision syndrome at the workplace. J Clin Epidemiol. 2015 Jun;68(6):662-73. doi: 10.1016/j.jclinepi.2015.01.015. Epub 2015 Jan 28. PMID 25744132
- [Background] Irmayani AI, Siregar AF, Lubis AS, Pratama MY, Lubis FH. Design and Trial of Computer Vision Syndrome Level Instruments.
- [Background] Kaiti R, Shah P, Bogati B, Shyangbo R, Dahal M, Hamal B. Computer vision syndrome: is it being diagnosed and managed properly. Acta Sci Ophthalmol. 2020;3(7):13-20.
- [Background] Abudawood GA, Ashi HM, Almarzouki NK. Computer vision syndrome among undergraduate medical students in King Abdulaziz University, Jeddah, Saudi Arabia. Journal of Ophthalmology. 2020 Apr 1;2020.
- [Background] Erdinest N, Berkow D. [COMPUTER VISION SYNDROME]. Harefuah. 2021 Jun;160(6):386-392. Hebrew. PMID 34160157
- [Background] Kang JI, Jeong DK, Park SK, Yang DJ, Kim JH, Moon YJ, Baek SY. Effect of Self-Stretching Exercises on Postural Improvement in Patients with Chronic Neck Pain Caused by Forward Head Posture. Journal of the Korean Society of Physical Medicine. 2020;15(3):51-9.